CLINICAL TRIAL: NCT03879122
Title: A Multi-arm, Multi-stage, Randomized Phase II/III Trial of Immunotherapy Strategies in Metastatic Hormone-sensitive Prostate Cancer
Brief Title: A Trial of Immunotherapy Strategies in Metastatic Hormone-sensitive Prostate Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Syntax for Science, S.L (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9HX
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
Keywords: prostate cancer; immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; Nivolumab; Docetaxel; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Multi-arm multi-stage (MAMS), multi-centre randomised controlled trial with 3 arms (2 experimental arms and a control arm) and 4 stages (three intermediate and a final stage). In all 3 intermediate stages of the trial, each experimental arm is compared in a pairwise manner with the control arm using an "intermediate" outcome measure. Experimental arms that do not reach a predefined critical value are discontinued. In the final stage, the remaining(s) arm(s) will be compared with the control arm in terms of overall survival (definitive outcome). The 3 arms included in this trial are the Control arm (ARM 1): ADT plus 6 cycles of DOCETAXEL and 2 experimental arms: ADT plus DOCETAXEL plus NIVOLUMAB (ARM 2) and ADT plus IPILIMUMAB alternating with DOCETAXEL and with NIVOLUMAB (ARM 3). Other experimental arms could be included later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADT + Docetaxel (Active Comparator): ADT (androgen deprivation therapy) plus 6 cycles of DOCETAXEL
  Interventions: Drug: Docetaxel; Drug: ADT (androgen deprivation therapy)
- ADT + Docetaxel + Nivolumab (Experimental): ADT (androgen deprivation therapy) plus DOCETAXEL plus NIVOLUMAB
  Interventions: Drug: Nivolumab 10 MG/ML; Drug: Docetaxel; Drug: ADT (androgen deprivation therapy)
- ADT + Ipilimumab / Docetaxel + Nivolumab (Experimental): ADT (androgen deprivation therapy) plus IPILIMUMAB alternating with DOCETAXEL and followed by NIVOLUMAB
  Interventions: Drug: Ipilimumab 5 MG/ML; Drug: Nivolumab 10 MG/ML; Drug: Docetaxel; Drug: ADT (androgen deprivation therapy)

INTERVENTIONS:
Drug: Ipilimumab 5 MG/ML — Ipilimumab will be administered on day 1 of each cycle every 3 weeks. In arm 3, ipilimumab should be started at least 2 weeks but no later than 120 days after surgical castration or the first dose of LHRH analogue. Patients should receive 2 doses of ipilimumab (6 weeks). It will be followed, 3 weeks later, by 3 cycles of docetaxel and by 2 additional doses of ipilimumab and 3 more cycles of docetaxel. Four weeks later, Nivolumab will be administered on day 1 every 2 weeks until a maximum of 24 doses (48 weeks)
  Other Names: YERVOY
  Arms: ADT + Ipilimumab / Docetaxel + Nivolumab
Drug: Nivolumab 10 MG/ML — Nivolumab will be administered every 2 weeks, until clinical progression or a maximum of 24 doses. Nivolumab should be started 4 weeks after the last dose of docetaxel, providing all the adverse effects have recovered, as if a new cycle of docetaxel were to be administered
  Other Names: Opdivo
  Arms: ADT + Docetaxel + Nivolumab; ADT + Ipilimumab / Docetaxel + Nivolumab
Drug: Docetaxel — Docetaxel should be given on day 1 every 21 days, for up to 6 cycles (1 cycle = 21 days). Docetaxel should be started within 7 working days from the date of randomization in the arm 1 and 2.
  In arm 3, docetaxel will be given 3 weeks after the last dose of the previous treatment, providing all the side effects are grade ≤1.
Drug: ADT (androgen deprivation therapy) — Androgen deprivation therapy per the standard of care

SUMMARY:
Metastatic prostate cancer is an incurable disease that typically spreads beyond the prostate. The standard of care is to systemically treat the disease with androgen deprivation therapy (ADT). However, the disease progresses in virtually all patients to the state of castration resistant prostate cancer (CRPC), with a median time to progression of 24 months. Patients with high volume disease (with either visceral metastasis and/or bone metastasis) exhibit a worse prognosis, with a median clinical progression of 14 months.

Recently, the CHAARTED and STAMPEDE studies demonstrated that the combination of Docetaxel (chemotherapy) and ADT delayed the clinical progression and improved the survival a median of 14 months (17 for high volume patients). Nevertheless, the prognosis of patients with high volume metastatic disease continues to be poor.

Meanwhile the immunotherapy, the use of antibodies that recognize tumoral cells and promote the immune system activity against the cancer, has emerged as a very useful option in many cancers. Among others, the antibodies Nivolumab and Ipilimumab have been approved for the treatment of multiple types of cancer.

In this context, SOGUG (Spanish Oncology Genitourinary Group) has designed this new study "PROSTRATEGY" with the objective of evaluating whether the addition of immunotherapy to chemotherapy and ADT improves the prognosis and survival of patients with high volume metastatic hormone-sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age
2. Signed and dated written informed consent, obtained before the performance of any protocol-related procedure.
3. Histological or cytological diagnosis of prostate cancer with an elevated PSA level and radiologic evidence of metastatic disease.
4. ECOG performance-status score of 0, 1, or 2. Patients with a score of 2 are eligible if the decrement in functioning was due to prostate cancer.
5. Metastatic disease that has spread beyond the prostate or relapsed after local therapy, documented by body CT scan and/or bone scan, according to PCWG 3 criteria, with high volume according to criteria used in the CHAARTED study.
6. Radiological and scintigraphic studies to identify initial evaluable disease should be done as follows:

   * If ADT has not been initiated, CT scans and bone scan must be obtained within 6 weeks prior to the start of ADT.
   * If all required imaging had not been completed prior to starting ADT, any additional scan must be obtained after starting androgen deprivation but prior to randomization and the initiation of docetaxel (It is assumed that the scans of patients with high volume disease would not normalize in less than 120 days to the point that a patient would go from "high volume" to "low volume").
7. Measurable or evaluable disease according to the PWGC 3.
8. Patients who started ADT for metastatic disease are eligible if ADT commenced within 120 days before randomization, they have not started docetaxel chemotherapy yet, and there was no evidence of clinical, radiological or biochemical progression after ADT.
9. Patients receiving ADT in the adjuvant and/or neoadjuvant setting for less than 30 months of therapy, AND the effect of the last depot injection had expired at least 12 months prior to documentation of metastatic disease, AND

   * They had no evidence of disease (PSA < 0.2 ng/dL) after prostatectomy plus hormonal therapy, or
   * PSA was < 0.5 ng/dL after completing radiation therapy plus adjuvant or neoadjuvant hormonal therapy, and had not doubled above nadir in at least 12 months.
10. Patients must have adequate organ function within 4 weeks prior to randomization and evidenced by:

    * Absolute Neutrophil Count > 1500/mm 3
    * Platelet count > 100,000/mm 3
    * Creatinine clearance (CrCl)> 30 mL/min calculated at screening using the Cockcroft- Gault formula: Creatinine clearance for mule (mL/min) = (140- age in years)(body weight in kg)/[72x(serum creatinine in mg/dl).
    * Total bilirubin < 1.5 ULN (< 3.0 mg/dl in patients with Gilbert´s Syndrome).
    * Prothrombin time or INR and PTT < 1.5 x ULN, except if on therapeutic anti- coagulation in which case the patient can be enrolled if stable and anti-coagulation levels are appropriate for their condition per good clinical practice.
    * ALT and AST < or = 3 x ULN (or < or = 5 if liver metastases)
11. At least 4 weeks should have passed after major surgery prior to randomization, and the patient should be recovered from all side effects and complications.
12. Men who are sexually active with WOCBP must agree to follow instructions for methods of contraception for the duration of treatment with study drug plus 5 half-lives of study drug plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion.

Exclusion Criteria:

1. Patients are not eligible if the PSA has risen from its lowest point, between the beginning of androgen deprivation therapy and the date of randomization, and met criteria for progression as defined in the protocol.
2. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, PROSTVAC, Sipuleucel-T or any previous immunotherapy or vaccines for cancer.
3. Prior chemotherapy in the adjuvant or neoadjuvant setting.
4. Unable to receive docetaxel at full doses at investigator criteria.
5. Peripheral neuropathy grade > 1.
6. All toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia or fatigue must have resolved to Grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. Subjects with toxicities attributed to prior surgery or radiotherapy, which are not expected to resolve and result in long-term lasting sequelae, are permitted to enrol.
7. History of hypersensitivity reaction to Docetaxel®, other drugs formulated with polysorbate 80, or monoclonal antibodies.
8. Prior hormone therapy or immunotherapy in the metastatic setting.
9. Prior palliative radiation therapy within 30 days of starting docetaxel.
10. Known acute or chronic HIV, Hepatitis B, or Hepatitis C. Past Hepatitis B infection with no signs of activity later, are allowed
11. Active brain metastases or leptomeningeal metastases, except if they have been treated and there is a magnetic resonance imaging (or CT scan if MRI were contraindicated) showing no evidence of progression for at least 4 weeks after the treatment
12. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days previous to randomization. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
13. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed.
14. Active cardiac disease defined as active angina, symptomatic congestive heart failure, or myocardial infarction within the previous six months
15. History of malignancy in the past 5 years except for basal cell and squamous cell carcinoma of the skin and non-muscle-invasive bladder cancer. Other more malignancies considered to have a low potential to progress may be enrolled if approved by study chair.
16. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
17. Participation in another clinical trial within 30 days prior to randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Condition is exclusive of males
Enrollment: 135 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 2 years
  Overall Survival

SECONDARY OUTCOMES:
PSA response | through study completion, an average of 2 years
PSA progression-free survival (PSA-PFS) | through study completion, an average of 2 years
Radiological progression-free survival (rPFS) | through study completion, an average of 2 years
Clinical progression-free survival (cPFS) | through study completion, an average of 2 years
Time to castration resistant prostate cancer (TCRPC) | through study completion, an average of 2 years
Immune radiological progression-free survival (irPFS) | through study completion, an average of 2 years
Immune clinical progression-free survival (icPFS) | through study completion, an average of 2 years
Time to immune castration resistant prostate cancer (TiCRPC) | through study completion, an average of 2 years
Symptomatic skeletal-related event free survival (SSREFS) | through study completion, an average of 2 years
Toxicity of each of the treatment arms by assessing Adverse Events | through study completion, an average of 2 years
Quality of life (QOL) | through study completion, an average of 2 years
  EQ-5D Questionnaire
Quality of life (QOL) | through study completion, an average of 2 years
  FACT-P Questionnaire
Quality of life (QOL) | through study completion, an average of 2 years
  BPI Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ángel Arranz Arija, MD, PhD, Principal Investigator — Physician - Investigator
Locations (30):
- Spain (30):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hestia Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sant Joan de Deu (Althaia Manresa), Manresa, Barcelona
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital General, Materno E Infantil Reina, Córdoba, Cordoba
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Arnau de Vilanova, Valencia, Valenci
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen Del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen de La Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Undecided